CLINICAL TRIAL: NCT02823665
Title: The Effects of Bariatric Surgeries on Glucose Metabolism
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 20180070H; 1R01DK105379-01 (NIH)
Record Dates: First submitted 2015-10-22; First posted 2016-07-06 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Post Bariatric Surgery; Gastric Bypass; Sleeve Gastrectomy; Hypoglycemia After Gastric Bypass
Keywords: gastric bypass surgery; Hypoglycemia; sleeve gastrectomy; glucose tolerance
MeSH Terms: conditions — Hypoglycemia | interventions — exendin (9-39); Atropine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exendin-(9-39) (Experimental): To evaluate the role of GLP-1 on glucose metabolism and insulin secretin after glucose and protein ingestion.
  Interventions: Drug: Exendin-(9-39)
- Atropine (Experimental): to evaluate the effect of neural activation on insulin secretion and glucose metabolism
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Exendin-(9-39) — A physiological study to evaluate the role of GLP-1 on glucose metabolism and insulin secretin after glucose and protein ingestion.
  Other Names: no other name for Exendin-(9-39)
  Arms: Exendin-(9-39)
Drug: Atropine — A physiological study to evaluate the effect of neural activation on insulin secretion and glucose metabolism.
  Other Names: Atropine sulfate
  Arms: Atropine

SUMMARY:
The purpose of this study is learn the effect of gastric bypass surgery and sleeve gastrectomy on glucose metabolism mediated by neural and hormonal factors initiated after eating.

DETAILED DESCRIPTION:
The purpose of this study is to determine the weight-independent effects of gastric bypass surgery and sleeve gastrectomy surgery on islet cell response after meal ingestion as mediated by hormonal and neural components of the gut. It will also address the differences between the two procedures.

Such information will be critical for the development of novel approaches for treatment of diabetes as well as improvement of glycemic effects of gastric bypass and sleeve gastrectomy in patients with partial diabetes remission or relapse after complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Hypoglycemic RYGB patients with documented blood glucose level <50 mg/dl
* Asymptomatic individuals with bariatric surgery
* Healthy non-surgical patients with no personal history of diabetes
* Subjects must physically be able to come to our clinical research center Cedars-Sinai Medical Center

Exclusion Criteria:

* Active heart, lung, liver, gastrointestinal or kidney disease; unable to give informed consent; pregnancy; uncontrolled high blood pressure or high cholesterol; significant anemia (hemoglobin <11g/dL); prisoners or institutionalized individuals; type 2 diabetes mellitis; development of any serious medical or psychiatric illness during recruitment or studies;
* RYGB patients will be disqualified if they have gastric outlet obstruction or severe diarrhea.
* Healthy non-surgical patients with personal history of diabetes

For administration of atropine, the following exclusions also apply:

* History of glaucoma
* Uncontrolled hypertension (any subjects with BP>140/90 and history of dyslipidemia
* Taking any medication that might interact with atropine and cannot be stopped will be excluded from the study)
* Myasthenia gravis
* Brain pathology
* Enlarged prostate in men

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Insulin levels measured after nutrient ingestion | Each study in the protocol is conducted up to seven hours with data collected at intervals specific to the individual study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Salehi, MD, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No